CLINICAL TRIAL: NCT02489344
Title: An Open-label, Multicenter, Multinational Extension Study of the Long-term Safety, Pharmacodynamics, and Exploratory Efficacy of GZ/SAR402671 in Adult Male Patients Diagnosed With Fabry Disease
Brief Title: Evaluation of the Long-term Safety, Pharmacodynamics, and Exploratory Efficacy of GZ/SAR402671 in Treatment-Naïve Adult Male Patients With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS14116; 2014-004995-49 (EudraCT Number); U1111-1165-9049 (Other: UTN)
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — venglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GZ/SAR402671 (Experimental): Participants received GZ/SAR402671 15 milligrams (mg) once daily orally for 30 months in this extension study (LTS14116).
  Interventions: Drug: GZ/SAR402671

INTERVENTIONS:
Drug: GZ/SAR402671 — Pharmaceutical form:capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

To assess the long-term safety of GZ/SAR402671 in adult male participants with Fabry disease who previously completed study ACT13739 (NCT02489344).

Secondary Objective:

To assess the long-term effect of GZ/SAR402671 on pharmacodynamic and exploratory efficacy endpoints in adult male participants with Fabry disease who previously completed study ACT13739.

DETAILED DESCRIPTION:
The total duration of this extension study (LTS14116) was up to 31 months (30 months of treatment and one month post-treatment follow-up).

ELIGIBILITY:
Inclusion criteria :

* Male participant with Fabry disease who previously completed study ACT13739.
* Participants, willing and able to provide signed informed consent.
* Sexually active participants, willing to practice true abstinence in line with their preferred and usual lifestyle or using two acceptable effective methods of contraception.

Exclusion criteria :

-Participants, in the opinion of the Investigator, unable to adhere to the requirements of the study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- United States (3):
  - Investigational Site Number 840002, Atlanta, Georgia
  - Investigational Site Number 840003, Cincinnati, Ohio
  - Investigational Site Number 840001, Fairfax, Virginia
- Investigational Site Number 250001, Garches, France
- Investigational Site Number 616001, Warsaw, Poland
- Investigational Site Number 643002, Moscow, Russia
- Investigational Site Number 826002, Cambridge, United Kingdom

REFERENCES:
- [Derived] Deegan PB, Goker-Alpan O, Geberhiwot T, Hopkin RJ, Lukina E, Tylki-Szymanska A, Zaher A, Sensinger C, Gaemers SJM, Modur V, Thurberg BL, Sharma J, Najafian B, Mauer M, DasMahapatra P, Wilcox WR, Germain DP. Venglustat, an orally administered glucosylceramide synthase inhibitor: Assessment over 3 years in adult males with classic Fabry disease in an open-label phase 2 study and its extension study. Mol Genet Metab. 2023 Feb;138(2):106963. doi: 10.1016/j.ymgme.2022.11.002. Epub 2022 Nov 9. PMID 36481125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who successfully completed 26 weeks of treatment in prior ACT13739 study (NCT02228460) were eligible to continue their treatment for up to 30 additional months in this extension study LTS14116. Eleven participants had enrolled and were treated in ACT13739 study, and 9 completed study. Of these 9 participants, 8 entered extension study.
Pre-assignment Details: In extension study, participants continued on same dose regimen they had received in initial study. Two participants in LTS14116 completed treatment and did not discontinue early, but are counted as not completed study due to no record of completion.
Groups:
- GZ/SAR402671: Participants received GZ/SAR402671 15 mg once daily orally for 36 months during combined ACT13739/LTS14116 treatment period.
Period: ACT13739 (Initial Study): 26 Weeks
Arm/Group | GZ/SAR402671
Started (Enrolled and treated.) | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Period: LTS14116 (Extension Study): 31 Months
Arm/Group | GZ/SAR402671
Started (Enrolled and treated.) | 8
Completed (2 participant completed,not discontinued early,but counted not completed due to no completion record) | 5
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Treatment completed/Study not completed | 2

BASELINE CHARACTERISTICS:
Population: Analysis performed on all participants who were initially enrolled in the ACT13739 study.
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian/White | 8
  Race: Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an adverse event (AE) without regard to possibility of causal relationship with this treatment. TEAEs were defined as AEs that developed or worsened during TEAE period (period from the first administration of study drug in ACT13739 through the last administration of the study drug in the combined ACT13739/LTS14116 treatment period plus 1 month or end of study participation for participant, whichever occurred first). For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: Analysis was performed on safety population: all participants who received at least 1 dose of investigational medicinal product (IMP) during the ACT13739 study. All data collected during ACT13739 and LTS14116 studies were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants | 9

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Hematological Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Hemoglobin: less than or equal to (<=) 115 grams per liter (g/L); greater than or equal to (>=)185 g/L; decreased from baseline (DFB) >=20 g/L
  * Hematocrit: <=0.37 volume/volume (v/v); >=0.55 v/v
  * Erythrocytes: >=6 Tera/L
  * Platelets: lesser than (<) 100 Giga/L; >=700 Giga/L
  * Leukocytes: <3.0 Giga/L (Non-Black [NB]) or <2.0 Giga/L (Black [B]); >=16.0 Giga/L
  * Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B);
  * Lymphocytes: greater than (>) 4.0 Giga/L
  * Monocytes: >0.7 Giga/L
  * Basophils: >0.1 Giga/L
  * Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L) For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: Analysis was performed on safety population: all participants who received at least 1 dose of IMP during the ACT13739 study. All data collected during ACT13739 and LTS14116 studies were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Hemoglobin <=115 g/L | 1
  Hemoglobin >=185 g/L | 0
  Hemoglobin DFB >=20 g/L | 0
  Hematocrit <=0.37 v/v | 6
  Hematocrit >0.55 v/v | 0
  Erythrocytes: >=6 Tera/L | 0
  Platelets <100 Giga/L | 0
  Platelets >=700 Giga/L | 0
  Leukocytes <3.0 Giga/L (NB) or <2.0 Giga/L (B) | 0
  Leukocytes >=16.0 Giga/L | 0
  Neutrophils <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 0
  Lymphocytes >4.0 Giga/L | 0
  Monocytes >0.7 Giga/L | 2
  Basophils >0.1 Giga/L | 1
  Eosinophils >0.5 Giga/L or >ULN (ULN >=0.5 Giga/L) | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Electrolytes
Description: Criteria for potentially clinically significant abnormalities:
  * Sodium: <=129 millimoles (mmol)/L; >=160 mmol/L
  * Potassium: <3 mmol/L; >=5.5 mmol/L
  * Chloride: <80 mmol/L; >115 mmol/L.
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Sodium <=129 mmol/L | 0
  Sodium >=160 mmol/L | 0
  Potassium <3 mmol/L | 0
  Potassium >=5.5 mmol/L | 0
  Chloride <80 mmol/L | 0
  Chloride >115 mmol/L | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Liver Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Alanine Aminotransferase (ALT): >3 ULN; >5 ULN; >10 ULN and >20 ULN
  * Aspartate aminotransferase (AST): >3 ULN; >5 ULN; >10 ULN and >20 ULN
  * Alkaline phosphatase: >1.5 ULN
  * Bilirubin: >1.5 ULN; >2 ULN.
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  ALT >3 ULN | 0
  ALT >5 ULN | 0
  ALT >10 ULN | 0
  ALT >20 ULN | 0
  AST >3 ULN | 0
  AST >5 ULN | 0
  AST >10 ULN | 0
  AST >20 ULN | 0
  Alkaline Phosphatase >1.5 ULN | 0
  Bilirubin >1.5 ULN | 0
  Bilirubin >2 ULN | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Metabolic Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Glucose: <=3.9 mmol/L and < lower limits of normal (LLN); >=11.1 mmol/L (unfasted [unfas]) or >=7 mmol/L (fasted [fas])
  * Lipase: >= 3 ULN
  * C Reactive Protein (CRP): > 2 ULN or > 10 milligrams (mg)/L (if ULN not provided).
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Glucose <=3.9 mmol/L and <LLN | 3
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas) | 1
  Albumin <=25 g/L | 0
  Lipase >=3 ULN | 0
  CRP >2 ULN or >10 mg/L (if ULN not provided) | 2

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Renal Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Creatinine: >=150 micromoles per liter (mcmol/L) (Adults); >=30% change from baseline; >= 100% change from baseline
  * Blood urea nitrogen: >=17 mmol/L
  * Urate: <120 mcmol/L; >408 mcmol/L For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Creatinine >=150 mcmol/L | 0
  Creatinine >=30% change from baseline | 2
  Creatinine >=100% change from baseline | 0
  Blood Urea Nitrogen >=17 mmol/L | 0
  Urate <120 mcmol/L | 0
  Urate >408 mcmol/L | 5

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Urinalysis
Description: Criteria with potentially clinically significant urine abnormalities:
  pH: <= 4.6; pH: >= 8.0
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  pH <= 4.6 | 0
  pH >= 8.0 | 0

8. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities:
  * Systolic blood pressure (SBP) supine: <=95 millimeters of mercury (mmHg) and DFB >=20 mmHg; >=160 mmHg and increase from baseline (IFB) >=20 mmHg
  * Diastolic blood pressure (DBP) supine: <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg
  * Heart rate (HR) supine: <=50 beats per minute (bpm) and DFB >=20 bpm; >=120 bpm and IFB >=20 bpm
  * Weight: >=5% DFB; >=5% IFB For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  SBP (supine) <=95 mmHg and DFB >=20 mmHg | 0
  SBP (supine) >=160 mmHg and IFB >=20 mmHg | 0
  DBP (supine) <=45 mmHg and DFB >=10 mmHg | 0
  DBP (supine) >=110 mmHg and IFB >=10 mmHg | 0
  HR (supine) <=50 bpm and DFB >= 20 bpm | 1
  HR (supine) >=120 bpm and IFB >=20 bpm | 0
  Weight >=5% DFB | 3
  Weight >=5% IFB | 2

9. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for potentially clinically significant ECG abnormalities:
  * ECG mean HR: <30 bpm; <30 bpm and DFB >=20 bpm; <40 bpm; <40 bpm and DFB >=20 bpm; <50 bpm; <50 bpm and DFB >=20 bpm; >90 bpm; <90 bpm and DFB >=20 bpm; >100 bpm; <100 bpm and DFB >=20 bpm; >120 bpm; <120 bpm and DFB >=20 bpm
  * PR Interval: >200 milliseconds (ms); >200 ms and IFB >=25%; >220 ms; >220 ms and IFB >=25%; >240 ms; >240 ms and IFB >=25%
  * QRS duration: >110 ms; >110 ms and IFB >=25%; >120 ms; >120 ms and IFB >=25%
  * QTc Bazett (QTcB) interval: >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms, IFB >60 ms
  * QTc Fridericia (QTc F): >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms; IFB >60 ms
  * QT Interval: >500 ms For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  ECG Mean HR <30 bpm | 0
  ECG Mean HR <30 bpm and DFB >=20 bpm | 0
  ECG Mean HR <40 bpm | 0
  ECG Mean HR <40 bpm and DFB >=20 bpm | 0
  ECG Mean HR <50 bpm | 1
  ECG Mean HR <50 bpm and DFB >=20 bpm | 0
  ECG Mean HR >90 bpm | 1
  ECG Mean HR <90 bpm and DFB >=20 bpm | 0
  ECG Mean HR >100 bpm | 0
  ECG Mean HR <100 bpm and DFB >=20 bpm | 0
  ECG Mean HR >120 bpm | 0
  ECG Mean HR <120 bpm and DFB >=20 bpm | 0
  PR interval >200 ms | 2
  PR interval >200 ms and IFB >=25% | 0
  PR interval >220 ms | 0
  PR interval >220 ms and IFB >=25% | 0
  PR >240 ms | 0
  PR interval >240 ms and IFB >=25% | 0
  QRS duration >110 ms | 1
  QRS duration >110 ms and IFB >=25% | 0
  QRS duration >120 ms | 0
  QRS duration >120 ms and IFB >=25% | 0
  QTcB interval >450 ms | 0
  QTcB interval >480 ms | 0
  QTc B interval >500 ms | 0
  QTcB interval IFB >30 and <=60 ms | 1
  QTcB interval IFB >60 ms | 0
  QTcF interval >450 ms | 0
  QTc F interval >480 ms | 0
  QTcF interval >500 ms | 0
  QTcF interval IFB >30 and <=60 ms | 0
  QTcF interval IFB >60 ms | 0
  QT interval >500 ms | 0

10. Secondary Outcome: Change From Baseline in Plasma Globotriaosylceramide (GL-3) Concentration at Weeks 26, 52, 104, and 156
Description: Change from baseline in plasma GL-3 was obtained by subtracting baseline value from post-baseline value at Weeks 26, 52, 104, and 156. Concentration of GL-3 in plasma was determined using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: Analysis was performed on full analysis set: all participants who received at least 1 dose of IMP during the ACT13739 study. All data collected during ACT13739 and LTS14116 studies were included in analysis. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
micrograms per milliliter (mcg/mL)
  Week 26: number analyzed (Participants) | 9
  Week 26 | -3.62 (1.07)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -5.06 (1.04)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -6.32 (2.53)
  Week 156: number analyzed (Participants) | 7
  Week 156 | -6.97 (2.27)

11. Secondary Outcome: Change From Baseline in Plasma Lyso Globotriaosylceramide (Lyso GL-3) Concentration at Weeks 26, 52, 104, and 156
Description: Change from baseline in plasma GL-3 was obtained by subtracting baseline value from post-baseline value at Weeks 26, 52, 104, and 156. Concentration of lyso-GL-3 in plasma was determined using a validated LC-MS/MS method. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nanograms per mL (ng/mL)
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
nanograms per mL (ng/mL)
  Week 26: number analyzed (Participants) | 9
  Week 26 | -30.99 (22.83)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -37.10 (20.69)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -39.84 (18.12)
  Week 156: number analyzed (Participants) | 7
  Week 156 | -48.13 (15.65)

12. Secondary Outcome: Change From Baseline in Plasma Glucosylceramide (GL-1) Concentration At Weeks 26, 52, 104, and 156
Description: Change from baseline in plasma GL-1 was obtained by subtracting baseline value from post-baseline value at Weeks 26, 52, 104, and 156. Concentration of GL-1 in plasma was determined using a validated LC-MS/MS method. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
mcg/mL
  Week 26: number analyzed (Participants) | 9
  Week 26 | -3.26 (1.43)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -3.58 (0.85)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -3.70 (0.85)
  Week 156: number analyzed (Participants) | 7
  Week 156 | -3.23 (1.11)

13. Secondary Outcome: Change From Baseline in Plasma Monosialodihexosylganglioside (GM3) Concentration At Weeks 26, 52, 104, and 156
Description: Change from baseline in plasma GM3 was obtained by subtracting baseline value from post-baseline value at Weeks 26, 52, 104, and 156. Concentration of GM3 in plasma was determined using a validated LC-MS/MS method. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
mcg/mL
  Week 26: number analyzed (Participants) | 9
  Week 26 | -10.77 (6.02)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -8.84 (4.55)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -9.92 (3.26)
  Week 156: number analyzed (Participants) | 7
  Week 156 | -8.12 (5.37)

14. Secondary Outcome: Change From Baseline in Urine GL-3 Concentration At Weeks 26, 52, 104, and 156
Description: Change from baseline in urine GL-3 was obtained by subtracting baseline value from post-baseline value at Weeks 26, 52, 104, and 156. Concentration of GL-3 in urine was determined using a validated LC-MS/MS method. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/mmol creatinine (Cr)
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
mg/mmol creatinine (Cr)
  Week 26: number analyzed (Participants) | 8
  Week 26 | -0.25 (0.19)
  Week 52: number analyzed (Participants) | 6
  Week 52 | -0.20 (0.22)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -0.18 (0.22)
  Week 156: number analyzed (Participants) | 7
  Week 156 | -0.18 (0.27)

15. Secondary Outcome: Change From Baseline in High Sensitivity Cardiac Troponin T At Weeks 26, 52, 104, and 156
Description: Change from baseline in high sensitivity cardiac troponin T was obtained by subtracting baseline value from post-baseline value at Weeks 26, 52, 104, and 156. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
mcg/L
  Week 26: number analyzed (Participants) | 9
  Week 26 | 0.0000 (0.0000)
  Week 52: number analyzed (Participants) | 5
  Week 52 | 0.0105 (0.0241)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -0.0015 (0.0000)
  Week 156: number analyzed (Participants) | 7
  Week 156 | 0.0006 (0.0027)

16. Secondary Outcome: Change From Baseline in Podocyturia Counts (Per Milligram of Creatinine) At Weeks 12, 26, and 156
Description: Change from baseline in podocyturia was obtained by subtracting baseline value from post-baseline value at Weeks 12, 26, and 156. Urine samples were processed to identify podocyte (podocalyxin, PCX) and parietal cell (claudin 1, CL1) markers. PCX +/CL1 negative cells were identified as podocytes and PCX +/CL1 positive cells as parietal cells with podocyte phenotype. All counts were corrected for urine Cr. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 12, 26, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Count of podocytes/mg Cr
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Count of podocytes/mg Cr
  Week 12: number analyzed (Participants) | 9
  Week 12 | -1.40 (2.69)
  Week 26: number analyzed (Participants) | 7
  Week 26 | -1.65 (2.97)
  Week 156: number analyzed (Participants) | 4
  Week 156 | -2.73 (3.97)

17. Secondary Outcome: Summary of Shifts From Baseline in Skin GL-3 Score in Superficial Capillary Endothelial Cells Over Time: Number of Participants in Categories of Shift in GL-3 Score
Description: Skin biopsies were performed for the scoring of GL-3 accumulation/inclusions by light microscopy. Three independent pathologists scored GL-3 clearance by using an inclusion severity score of 0 (none/trace), 1 (mild), 2 (moderate), and 3 (severe), where higher score indicated more severe condition. A single score per participant per time point was derived by taking the score rated by a majority of the pathologists; if a majority score could not be derived, the median score was used. Data were summarized and reported in terms of number of participants with shift from baseline GL-3 score to Weeks 12, 26, 52, and 156 GL-3 score. Shift to lower score from baseline indicated less severe condition at that respective time point. Any shift category of Baseline score/Week score that was not observed (no participant had data in the category) was not reported. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 12, 26, 52, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline Score:1/Week 12 Score:1: number analyzed (Participants) | 9
  Baseline Score:1/Week 12 Score:1 | 4
  Baseline Score:1/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:1/Week 12 Score:2 | 1
  Baseline Score:2/Week 12 Score:1: number analyzed (Participants) | 9
  Baseline Score:2/Week 12 Score:1 | 3
  Baseline Score:2/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 12 Score:2 | 1
  Baseline Score:1/Week 26 Score:1: number analyzed (Participants) | 9
  Baseline Score:1/Week 26 Score:1 | 4
  Baseline Score:1/Week 26 Score:2: number analyzed (Participants) | 9
  Baseline Score:1/Week 26 Score:2 | 1
  Baseline Score:2/Week 26 Score:1: number analyzed (Participants) | 9
  Baseline Score:2/Week 26 Score:1 | 3
  Baseline Score:2/Week 26 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 26 Score:2 | 1
  Baseline Score:1/Week 52 Score:1: number analyzed (Participants) | 6
  Baseline Score:1/Week 52 Score:1 | 3
  Baseline Score:2/Week 52 Score:1: number analyzed (Participants) | 6
  Baseline Score:2/Week 52 Score:1 | 2
  Baseline Score:2/Week 52 Score:2: number analyzed (Participants) | 6
  Baseline Score:2/Week 52 Score:2 | 1
  Baseline Score:1/Week 156 Score:0: number analyzed (Participants) | 6
  Baseline Score:1/Week 156 Score:0 | 2
  Baseline Sore:1/Week 156 Score:1: number analyzed (Participants) | 6
  Baseline Sore:1/Week 156 Score:1 | 1
  Baseline Score:2/Week 156 Score:1: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:1 | 3

18. Secondary Outcome: Summary of Shifts From Baseline in Skin GL-3 Score in Deep Vessels Endothelial Cells Over Time: Number of Participants in Categories of Shift in GL-3 Score
Description: as for outcome 17
Time Frame: Baseline of ACT13739 study and Weeks 12, 26, 52, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline Score:1/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:1/Week 12 Score:2 | 1
  Baseline Score:2/Week 12 Score:1: number analyzed (Participants) | 9
  Baseline Score:2/Week 12 Score:1 | 2
  Baseline Score:2/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 12 Score:2 | 6
  Baseline Score:1/Week 26 Score:1: number analyzed (Participants) | 9
  Baseline Score:1/Week 26 Score:1 | 1
  Baseline Score:2/Week 26 Score:1: number analyzed (Participants) | 9
  Baseline Score:2/Week 26 Score:1 | 2
  Baseline Score:2/Week 26 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 26 Score:2 | 6
  Baseline Score:2/Week 52 Score:1: number analyzed (Participants) | 6
  Baseline Score:2/Week 52 Score:1 | 3
  Baseline Score:2/Week 52 Score:1.5: number analyzed (Participants) | 6
  Baseline Score:2/Week 52 Score:1.5 | 1
  Baseline Sore:2/Week 52 Score:2: number analyzed (Participants) | 6
  Baseline Sore:2/Week 52 Score:2 | 2
  Baseline Score:1/Week 156 Score:1: number analyzed (Participants) | 6
  Baseline Score:1/Week 156 Score:1 | 1
  Baseline Score:2/Week 156 Score:0.5: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:0.5 | 1
  Baseline Score:2/Week 156 Score:1: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:1 | 3
  Baseline Score:2/Week 156 Score:2: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:2 | 1

19. Secondary Outcome: Summary of Shifts From Baseline in Skin GL-3 Score in Deep Vessels Smooth Muscle Cells Over Time: Number of Participants in Categories of Shift in GL-3 Score
Description: as for outcome 17
Time Frame: Baseline of ACT13739 study and Weeks 12, 26, 52, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline Score:1.5/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:1.5/Week 12 Score:2 | 2
  Baseline Score:2/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 12 Score:2 | 7
  Baseline Score:1.5/Week 26 Score:1.5: number analyzed (Participants) | 9
  Baseline Score:1.5/Week 26 Score:1.5 | 2
  Baseline Score:2/Week 26 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 26 Score:2 | 7
  Baseline Score:1.5/Week 52 Score:2: number analyzed (Participants) | 5
  Baseline Score:1.5/Week 52 Score:2 | 1
  Baseline Score:2/Week 52 Score:2: number analyzed (Participants) | 5
  Baseline Score:2/Week 52 Score:2 | 4
  Baseline Score:1.5/Week 156 Score:2: number analyzed (Participants) | 6
  Baseline Score:1.5/Week 156 Score:2 | 1
  Baseline Score:2/Week 156 Score:1: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:1 | 1
  Baseline Score:2/Week 156 Score:1.5: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:1.5 | 1
  Baseline Score:2/Week 156 Score:2: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:2 | 3

20. Secondary Outcome: Summary of Shifts From Baseline in Skin GL-3 Score in Perineurium Cells Over Time: Number of Participants in Categories of Shift in GL-3 Score
Description: as for outcome 17
Time Frame: Baseline of ACT13739 study and Weeks 12, 26, 52, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline Score:1/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:1/Week 12 Score:2 | 1
  Baseline Score:2/Week 12 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 12 Score:2 | 8
  Baseline Score:1/Week 26 Score:2: number analyzed (Participants) | 9
  Baseline Score:1/Week 26 Score:2 | 1
  Baseline Score:2/Week 26 Score:2: number analyzed (Participants) | 9
  Baseline Score:2/Week 26 Score:2 | 8
  Baseline Score:1/Week 52 Score:2: number analyzed (Participants) | 6
  Baseline Score:1/Week 52 Score:2 | 1
  Baseline Score:2/Week 52 Score:1: number analyzed (Participants) | 6
  Baseline Score:2/Week 52 Score:1 | 1
  Baseline Score:2/Week 52 Score:1.5: number analyzed (Participants) | 6
  Baseline Score:2/Week 52 Score:1.5 | 1
  Baseline Score:2/Week 52 Score:2: number analyzed (Participants) | 6
  Baseline Score:2/Week 52 Score:2 | 3
  Baseline Score:1/Week 156 Score:1: number analyzed (Participants) | 6
  Baseline Score:1/Week 156 Score:1 | 1
  Baseline Score:2/Week 156 Score:1.5: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:1.5 | 1
  Baseline Score:2/Week 156 Score:2: number analyzed (Participants) | 6
  Baseline Score:2/Week 156 Score:2 | 4

21. Secondary Outcome: Change From Baseline in Mental Component Summary and Physical Component Summary of the Short Form-36 (SF-36) Health Survey at Weeks 26, 52, 104 and 156
Description: The SF-36 health survey is a participant-reported survey to measure participant's health. It is a 36-item questionnaire used to measure 8 various aspects of health (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health). The score range for each of the 8 aspects was from 0 (maximum disability) to 100 (no disability), higher scores indicating good health condition. Responses on the SF-36 were also used to calculate 2 summary scores: Physical component score (PCS) and mental component score (MCS). The score range for each of these 2 summary scores was from 0 (maximum disability) to 100 (no disability), where higher score indicated less disability or good health condition. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
units on a scale
  Physical Component Summary: Week 26: number analyzed (Participants) | 9
  Physical Component Summary: Week 26 | 8.39 (6.88)
  Physical Component Summary: Week 52: number analyzed (Participants) | 7
  Physical Component Summary: Week 52 | 7.70 (7.76)
  Physical Component Summary: Week 104: number analyzed (Participants) | 6
  Physical Component Summary: Week 104 | 9.72 (9.02)
  Physical Component Summary: Week 156: number analyzed (Participants) | 6
  Physical Component Summary: Week 156 | 5.30 (11.83)
  Mental Component Summary: Week 26: number analyzed (Participants) | 9
  Mental Component Summary: Week 26 | -3.31 (20.34)
  Mental Component Summary: Week 52: number analyzed (Participants) | 7
  Mental Component Summary: Week 52 | 1.69 (8.27)
  Mental Component Summary: Week 104: number analyzed (Participants) | 6
  Mental Component Summary: Week 104 | 6.48 (8.14)
  Mental Component Summary: Week 156: number analyzed (Participants) | 6
  Mental Component Summary: Week 156 | 2.87 (14.17)

22. Secondary Outcome: Gastrointestinal (GI) Symptoms: Number of Participants With Abdominal Pain at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to report the presence of abdominal pain in past 10 days (before each of the specified time points). Participants answered the question: "Do you currently suffer from abdominal (tummy) pain? [Yes/No]". For this analysis, baseline was defined as initial ACT13739 study.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline: No | 5
  Baseline: Yes | 6
  Week 2: No | 6
  Week 2: Yes | 5
  Week 4: No | 7
  Week 4: Yes | 4
  Week 8: No | 8
  Week 8: Yes | 3
  Week 12: number analyzed (Participants) | 10
  Week 12: No | 8
  Week 12: Yes | 2
  Week 18: number analyzed (Participants) | 9
  Week 18: No | 7
  Week 18: Yes | 2
  Week 26: number analyzed (Participants) | 9
  Week 26: No | 6
  Week 26: Yes | 3
  Week 52: number analyzed (Participants) | 7
  Week 52: No | 5
  Week 52: Yes | 2
  Week 104: number analyzed (Participants) | 7
  Week 104: No | 5
  Week 104: Yes | 2
  Week 156: number analyzed (Participants) | 7
  Week 156: No | 5
  Week 156: Yes | 2

23. Secondary Outcome: Gastrointestinal Symptoms: Abdominal Pain Severity Score at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to mark the severity of the abdominal pain in past 10 days (before each of the specified time points) on a visual analogue scale (VAS). The scale ranged from 0% (no pain) to 100% (very severe), where higher score indicated more severity. For this analysis, baseline was defined as initial ACT13739 study baseline. Standard deviation (SD) can only be calculated when there are more than 1 participant with data available. Thereby, applicable fields were left blank when SD was not calculable.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a 0-100 percent scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
score on a 0-100 percent scale
  Baseline: number analyzed (Participants) | 6
  Baseline | 52.50 (20.50)
  Week 2: number analyzed (Participants) | 5
  Week 2 | 35.60 (18.47)
  Week 4: number analyzed (Participants) | 4
  Week 4 | 29.75 (20.07)
  Week 8: number analyzed (Participants) | 3
  Week 8 | 29.00 (21.28)
  Week 12: number analyzed (Participants) | 2
  Week 12 | 40.00 (21.21)
  Week 18: number analyzed (Participants) | 2
  Week 18 | 43.00 (29.70)
  Week 26: number analyzed (Participants) | 3
  Week 26 | 31.33 (32.81)
  Week 52: number analyzed (Participants) | 1
  Week 52 | 21.00
  Week 104: number analyzed (Participants) | 1
  Week 104 | 21.00
  Week 156: number analyzed (Participants) | 2
  Week 156 | 15.00 (7.07)

24. Secondary Outcome: Gastrointestinal Symptoms: Number of Days With Abdominal Pain Score at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to report the number of days they had abdominal pain in past 10 days (before each of the specified time points). Number of days with abdominal pain score was achieved by multiplying number of days with pain * 10. The score ranges from 10 to 100, where higher score signifies more number of days with pain. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
score on a scale
  Baseline: number analyzed (Participants) | 6
  Baseline | 38.33 (31.89)
  Week 2: number analyzed (Participants) | 5
  Week 2 | 26.00 (20.74)
  Week 4: number analyzed (Participants) | 4
  Week 4 | 25.00 (20.82)
  Week 8: number analyzed (Participants) | 4
  Week 8 | 25.00 (23.80)
  Week 12: number analyzed (Participants) | 2
  Week 12 | 35.00 (7.07)
  Week 18: number analyzed (Participants) | 2
  Week 18 | 35.00 (21.21)
  Week 26: number analyzed (Participants) | 3
  Week 26 | 30.00 (34.64)
  Week 52: number analyzed (Participants) | 3
  Week 52 | 7.00 (12.12)
  Week 104: number analyzed (Participants) | 2
  Week 104 | 5.00 (7.07)
  Week 156: number analyzed (Participants) | 2
  Week 156 | 20.00 (0.00)

25. Secondary Outcome: Gastrointestinal Symptoms: Number of Participants With Abdominal Distension at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to report the presence of abdominal distention in past 10 days (before each of the specified time points). Participants answered the question: "Do you currently suffer from abdominal distension (bloating, swelling or tight tummy)? [Yes/No]". For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline: No | 9
  Baseline: Yes | 2
  Week 2: No | 8
  Week 2: Yes | 3
  Week 4: No | 7
  Week 4: Yes | 4
  Week 8: No | 9
  Week 8: Yes | 2
  Week 12: number analyzed (Participants) | 10
  Week 12: No | 9
  Week 12: Yes | 1
  Week 18: number analyzed (Participants) | 9
  Week 18: No | 8
  Week 18: Yes | 1
  Week 26: number analyzed (Participants) | 9
  Week 26: No | 8
  Week 26: Yes | 1
  Week 52: number analyzed (Participants) | 7
  Week 52: No | 7
  Week 52: Yes | 0
  Week 104: number analyzed (Participants) | 7
  Week 104: No | 7
  Week 104: Yes | 0
  Week 156: number analyzed (Participants) | 7
  Week 156: No | 6
  Week 156: Yes | 1

26. Secondary Outcome: Gastrointestinal Symptoms: Abdominal Distension Severity Score at Baseline and Weeks 2, 4, 8, 12, 18, 26, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to mark the severity of the abdominal distension in past 10 days (before each of the specified time points) on a VAS. The scale ranged from 0% (no distention) to 100% (very severe), where higher score indicated more severity. For this analysis, baseline was defined as initial ACT13739 study baseline. The SD can only be calculated when there are more than 1 participant with data available. Thereby, applicable fields were left blank when SD was not calculable.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a 0-100 percent scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
score on a 0-100 percent scale
  Baseline: number analyzed (Participants) | 3
  Baseline | 45.33 (24.01)
  Week 2: number analyzed (Participants) | 3
  Week 2 | 38.67 (38.42)
  Week 4: number analyzed (Participants) | 4
  Week 4 | 21.00 (26.15)
  Week 8: number analyzed (Participants) | 2
  Week 8 | 35.00 (48.08)
  Week 12: number analyzed (Participants) | 1
  Week 12 | 72.00
  Week 18: number analyzed (Participants) | 1
  Week 18 | 69.00
  Week 26: number analyzed (Participants) | 1
  Week 26 | 80.00
  Week 156: number analyzed (Participants) | 1
  Week 156 | 5.00

27. Secondary Outcome: Gastrointestinal Symptoms: Number of Participants in Categories of Response Regarding Eating Less Due to Abdominal Pain/Bloating at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants responded to question "How often do you eat less during meals due to abdominal pain and/or bloating?" in past 10 days (before each of the specified time points) in the categories as 'never', 'occasionally' or 'often'. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline: Never | 4
  Baseline: Occasionally | 5
  Baseline: Often | 2
  Week 2: Never | 6
  Week 2: Occasionally | 3
  Week 2: Often | 2
  Week 4: Never | 6
  Week 4: Occasionally | 3
  Week 4: Often | 2
  Week 8: Never | 7
  Week 8: Occasionally | 3
  Week 8: Often | 1
  Week 12: number analyzed (Participants) | 10
  Week 12: Never | 5
  Week 12: Occasionally | 3
  Week 12: Often | 2
  Week 18: number analyzed (Participants) | 9
  Week 18: Never | 4
  Week 18: Occasionally | 3
  Week 18: Often | 2
  Week 26: number analyzed (Participants) | 9
  Week 26: Never | 4
  Week 26: Occasionally | 3
  Week 26: Often | 2
  Week 52: number analyzed (Participants) | 7
  Week 52: Never | 3
  Week 52: Occasionally | 3
  Week 52: Often | 1
  Week 104: number analyzed (Participants) | 7
  Week 104: Never | 4
  Week 104: Occasionally | 3
  Week 104: Often | 0
  Week 156: number analyzed (Participants) | 7
  Week 156: Never | 4
  Week 156: Occasionally | 3
  Week 156: Often | 0

28. Secondary Outcome: Gastrointestinal Symptoms: Satisfaction Over Bowel Habits at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to mark their satisfaction over bowel habits in past 10 days (before each of the specified time points) on a VAS. The scale ranged from 0% (very happy) to 100% (very unhappy), where higher percentage indicated less satisfaction. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a 0-100 percent scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
score on a 0-100 percent scale
  Baseline | 26.55 (19.09)
  Week 2 | 30.82 (21.17)
  Week 4 | 36.09 (28.68)
  Week 8 | 34.27 (27.02)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 21.50 (17.83)
  Week 18: number analyzed (Participants) | 9
  Week 18 | 23.89 (21.29)
  Week 26: number analyzed (Participants) | 9
  Week 26 | 35.56 (29.37)
  Week 52: number analyzed (Participants) | 6
  Week 52 | 19.00 (17.05)
  Week 104: number analyzed (Participants) | 5
  Week 104 | 18.00 (15.18)
  Week 156: number analyzed (Participants) | 6
  Week 156 | 34.02 (36.67)

29. Secondary Outcome: Gastrointestinal Symptoms: Frequency of Bowel Movements - Most Number of Times Bowel Movement Per Day at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to report the frequency of their bowel movement (per day or per week or per month) in past 10 days (before each of the specified time points) by answering the question "What is the most number of times you move your bowels per day/week/month?". Participants selected their preferred time unit (e.g., per day). Response provided by participants was converted to number of times per day for reporting the results. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: number of bowel movements per day
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
number of bowel movements per day
  Baseline | 2.36 (1.03)
  Week 2 | 2.00 (0.63)
  Week 4 | 2.00 (1.00)
  Week 8 | 1.74 (1.07)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 2.04 (1.08)
  Week 18: number analyzed (Participants) | 9
  Week 18 | 2.17 (1.05)
  Week 26: number analyzed (Participants) | 9
  Week 26 | 2.16 (1.07)
  Week 52: number analyzed (Participants) | 7
  Week 52 | 2.08 (1.00)
  Week 104: number analyzed (Participants) | 7
  Week 104 | 1.96 (1.05)
  Week 156: number analyzed (Participants) | 7
  Week 156 | 1.65 (0.61)

30. Secondary Outcome: Gastrointestinal Symptoms: Frequency of Bowel Movements - Least Number of Times Bowel Movement Per Day at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to report the frequency of their bowel movement (per day or per week or per month) in past 10 days (before each of the specified time points). Participants answered the question "What is the least number of times you move your bowels per day/week/month?". Participants selected their preferred time unit (e.g., per day). Response provided by participants was converted to number of times per day for reporting the results. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: number of bowel movements per day
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
number of bowel movements per day
  Baseline | 0.78 (0.56)
  Week 2 | 0.66 (0.43)
  Week 4 | 0.65 (0.62)
  Week 8 | 0.62 (0.64)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 0.67 (0.65)
  Week 18: number analyzed (Participants) | 9
  Week 18 | 0.73 (0.65)
  Week 26: number analyzed (Participants) | 9
  Week 26 | 0.75 (0.40)
  Week 52: number analyzed (Participants) | 7
  Week 52 | 0.76 (0.72)
  Week 104: number analyzed (Participants) | 7
  Week 104 | 0.61 (0.49)
  Week 156: number analyzed (Participants) | 7
  Week 156 | 0.92 (0.62)

31. Secondary Outcome: Gastrointestinal Symptoms: Influence of GI Symptoms of Fabry Disease on Life at Baseline and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156
Description: Participants assessed their GI symptoms (abdominal pain, abdominal distention, bowel movements) by completing a questionnaire (modified version of the inflammatory bowel severity scoring system). Participants were asked to mark the influence of their GI symptoms of Fabry disease on life in past 10 days (before each of the specified time points) on a VAS. The scale ranged from 0% (no at all) to 100% (completely), where higher percentage indicated more influence of the GI symptoms of the disease on life. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 2, 4, 8, 12, 18, 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a 0-100 percent scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
score on a 0-100 percent scale
  Baseline | 34.36 (26.47)
  Week 2 | 26.73 (25.22)
  Week 4 | 21.27 (19.88)
  Week 8 | 22.09 (19.77)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 17.50 (19.92)
  Week 18: number analyzed (Participants) | 9
  Week 18 | 24.89 (23.34)
  Week 26: number analyzed (Participants) | 9
  Week 26 | 36.44 (30.18)
  Week 52: number analyzed (Participants) | 6
  Week 52 | 20.33 (22.04)
  Week 104: number analyzed (Participants) | 5
  Week 104 | 26.50 (23.31)
  Week 156: number analyzed (Participants) | 6
  Week 156 | 19.82 (21.14)

32. Secondary Outcome: Gastrointestinal Symptoms: Number of Participants With Stool Consistency Assessment by Bristol Stool Scale Scoring at Baseline and Weeks 26, 52, 104, and 156
Description: Participants were asked to rate their stool consistency in past 10 days (before each of the specified time points) on a 7-point Bristol stool scale, according to the following types: 1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = sausage-like with cracks on the surface, 4 = sausage-like but smooth and soft, 5 = soft blobs with clear cut edges, 6 = fluffy pieces with ragged edges, and 7 = watery with no solid pieces. Types 1 and 2 indicate constipation, types 3 and 4 indicate "ideal stools" (easiest to defecate), and 5-7 tending towards diarrhea. Frequency of each stool type was categorized as 'never', occasionally', or 'often'. For this analysis, baseline was defined as the initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Stool Type 1: Baseline: Never | 11
  Stool Type 1: Baseline: Occasionally | 0
  Stool Type 1: Baseline: Often | 0
  Stool Type 1: Week 26: number analyzed (Participants) | 9
  Stool Type 1: Week 26: Never | 8
  Stool Type 1: Week 26: Occasionally | 1
  Stool Type 1: Week 26: Often | 0
  Stool Type 1: Week 52: number analyzed (Participants) | 7
  Stool Type 1: Week 52: Never | 6
  Stool Type 1: Week 52: Occasionally | 0
  Stool Type 1: Week 52: Often | 1
  Stool Type 1: Week 104: number analyzed (Participants) | 7
  Stool Type 1: Week 104: Never | 6
  Stool Type 1: Week 104: Occasionally | 0
  Stool Type 1: Week 104: Often | 1
  Stool Type 1: Week 156: number analyzed (Participants) | 7
  Stool Type 1: Week 156: Never | 5
  Stool Type 1: Week 156: Occasionally | 1
  Stool Type 1: Week 156: Often | 1
  Stool Type 2: Baseline: Never | 6
  Stool Type 2: Baseline: Occasionally | 5
  Stool Type 2: Baseline: Often | 0
  Stool Type 2: Week 26: number analyzed (Participants) | 9
  Stool Type 2: Week 26: Never | 6
  Stool Type 2: Week 26: Occasionally | 0
  Stool Type 2: Week 26: Often | 3
  Stool Type 2: Week 52: number analyzed (Participants) | 7
  Stool Type 2: Week 52: Never | 3
  Stool Type 2: Week 52: Occasionally | 4
  Stool Type 2: Week 52: Often | 0
  Stool Type 2: Week 104: number analyzed (Participants) | 7
  Stool Type 2: Week 104: Never | 4
  Stool Type 2: Week 104: Occasionally | 2
  Stool Type 2: Week 104: Often | 1
  Stool Type 2: Week 156: number analyzed (Participants) | 7
  Stool Type 2: Week 156: Never | 2
  Stool Type 2: Week 156: Occasionally | 3
  Stool Type 2: Week 156: Often | 2
  Stool Type 3: Baseline: Never | 1
  Stool Type 3: Baseline: Occasionally | 4
  Stool Type 3: Baseline: Often | 6
  Stool Type 3: Week 26: number analyzed (Participants) | 9
  Stool Type 3: Week 26: Never | 1
  Stool Type 3: Week 26: Occasionally | 3
  Stool Type 3: Week 26: Often | 5
  Stool Type 3: Week 52: number analyzed (Participants) | 7
  Stool Type 3: Week 52: Never | 0
  Stool Type 3: Week 52: Occasionally | 3
  Stool Type 3: Week 52: Often | 4
  Stool Type 3: Week 104: number analyzed (Participants) | 7
  Stool Type 3: Week 104: Never | 0
  Stool Type 3: Week 104: Occasionally | 6
  Stool Type 3: Week 104: Often | 1
  Stool Type 3: Week 156: number analyzed (Participants) | 7
  Stool Type 3: Week 156: Never | 0
  Stool Type 3: Week 156: Occasionally | 4
  Stool Type 3: Week 156: Often | 3
  Stool Type 4: Baseline: Never | 1
  Stool Type 4: Baseline: Occasionally | 8
  Stool Type 4: Baseline: Often | 2
  Stool Type 4: Week 26: number analyzed (Participants) | 9
  Stool Type 4: Week 26: Never | 2
  Stool Type 4: Week 26: Occasionally | 4
  Stool Type 4: Week 26: Often | 3
  Stool Type 4: Week 52: number analyzed (Participants) | 7
  Stool Type 4: Week 52: Never | 3
  Stool Type 4: Week 52: Occasionally | 1
  Stool Type 4: Week 52: Often | 3
  Stool Type 4: Week 104: number analyzed (Participants) | 7
  Stool Type 4: Week 104: Never | 2
  Stool Type 4: Week 104: Occasionally | 3
  Stool Type 4: Week 104: Often | 2
  Stool Type 4: Week 156: number analyzed (Participants) | 7
  Stool Type 4: Week 156: Never | 3
  Stool Type 4: Week 156: Occasionally | 2
  Stool Type 4: Week 156: Often | 2
  Stool type 5: Baseline: Never | 1
  Stool type 5: Baseline: Occasionally | 9
  Stool type 5: Baseline: Often | 1
  Stool type 5: Week 26: number analyzed (Participants) | 9
  Stool type 5: Week 26: Never | 4
  Stool type 5: Week 26: Occasionally | 4
  Stool type 5: Week 26: Often | 1
  Stool type 5: Week 52: number analyzed (Participants) | 7
  Stool type 5: Week 52: Never | 5
  Stool type 5: Week 52: Occasionally | 2
  Stool type 5: Week 52: Often | 0
  Stool type 5: Week 104: number analyzed (Participants) | 7
  Stool type 5: Week 104: Never | 4
  Stool type 5: Week 104: Occasionally | 1
  Stool type 5: Week 104: Often | 2
  Stool type 5: Week 156: number analyzed (Participants) | 7
  Stool type 5: Week 156: Never | 3
  Stool type 5: Week 156: Occasionally | 3
  Stool type 5: Week 156: Often | 1
  Stool Type 6: Baseline: Never | 5
  Stool Type 6: Baseline: Occasionally | 5
  Stool Type 6: Baseline: Often | 1
  Stool Type 6: Week 26: number analyzed (Participants) | 9
  Stool Type 6: Week 26: Never | 4
  Stool Type 6: Week 26: Occasionally | 4
  Stool Type 6: Week 26: Often | 1
  Stool Type 6: Week 52: number analyzed (Participants) | 7
  Stool Type 6: Week 52: Never | 4
  Stool Type 6: Week 52: Occasionally | 2
  Stool Type 6: Week 52: Often | 1
  Stool Type 6: Week 104: number analyzed (Participants) | 7
  Stool Type 6: Week 104: Never | 3
  Stool Type 6: Week 104: Occasionally | 3
  Stool Type 6: Week 104: Often | 1
  Stool Type 6: Week 156: number analyzed (Participants) | 7
  Stool Type 6: Week 156: Never | 4
  Stool Type 6: Week 156: Occasionally | 3
  Stool Type 6: Week 156: Often | 0
  Stool Type 7: Baseline: Never | 5
  Stool Type 7: Baseline: Occasionally | 5
  Stool Type 7: Baseline: Often | 1
  Stool Type 7: Week 26: number analyzed (Participants) | 9
  Stool Type 7: Week 26: Never | 5
  Stool Type 7: Week 26: Occasionally | 4
  Stool Type 7: Week 26: Often | 0
  Stool Type 7: Week 52: number analyzed (Participants) | 7
  Stool Type 7: Week 52: Never | 5
  Stool Type 7: Week 52: Occasionally | 2
  Stool Type 7: Week 52: Often | 0
  Stool Type 7: Week 104: number analyzed (Participants) | 7
  Stool Type 7: Week 104: Never | 4
  Stool Type 7: Week 104: Occasionally | 3
  Stool Type 7: Week 104: Often | 0
  Stool Type 7: Week 156: number analyzed (Participants) | 7
  Stool Type 7: Week 156: Never | 3
  Stool Type 7: Week 156: Occasionally | 3
  Stool Type 7: Week 156: Often | 1

33. Secondary Outcome: Change From Baseline in Beck Depression Inventory (BDI) Total Score at Weeks 26, 104, and 156
Description: The BDI-II Scale was a 21-item scoring tool which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represent a depressive symptom. Each symptoms were scored on a 4-point scale of 0 to 3 (0=symptom not present); (3=symptom very intense). Scores for each symptom were added up to obtain the total scores for all 21 items, which were interpreted as follows: Scores of 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression and 29-63: severe depression, where higher scores indicated more depression. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
score on a scale
  Week 26: number analyzed (Participants) | 9
  Week 26 | -0.89 (8.13)
  Week 104: number analyzed (Participants) | 4
  Week 104 | 2.00 (3.37)
  Week 156: number analyzed (Participants) | 7
  Week 156 | -3.43 (7.09)

34. Secondary Outcome: Change From Baseline in Albumin/Creatinine Ratio (ACR) and Protein/Creatinine Ratio (PCR) at Weeks 26, 52, 104, and 156
Description: For each scheduled visit for this assessment, 3 timed overnight urine samples were collected between 4 to 7 days of each other. All urine samples were collected within a 16-day period. ACR and PCR were determined for each collection. The median of the values determined for the 3 collections/visit was used for analysis. Baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
mg/g
  ACR: Week 26: number analyzed (Participants) | 9
  ACR: Week 26 | -26.22 (26.75)
  ACR: Week 52: number analyzed (Participants) | 7
  ACR: Week 52 | 1.00 (57.23)
  ACR: Week 104: number analyzed (Participants) | 7
  ACR: Week 104 | 12.21 (71.82)
  ACR: Week 156: number analyzed (Participants) | 7
  ACR: Week 156 | -1.14 (54.80)
  PCR: Week 26: number analyzed (Participants) | 9
  PCR: Week 26 | -38.33 (24.40)
  PCR: Week 52: number analyzed (Participants) | 7
  PCR: Week 52 | 0.33 (62.11)
  PCR: Week 104: number analyzed (Participants) | 7
  PCR: Week 104 | -12.88 (76.97)
  PCR: Week 156: number analyzed (Participants) | 7
  PCR: Week 156 | -34.38 (71.40)

35. Secondary Outcome: Number of Participants in Categories of Echocardiogram (ECHO) Results at Baseline and at Weeks 26, 52, 104, and 156
Description: The summary statistics of all continuous echocardiogram variables were calculated for each visit. The overall interpretation of the readings were summarized in 3 categories: normal, abnormal but not clinically significant (NCS), and abnormal but clinically significant (CS) categories. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline: number analyzed (Participants) | 8
  Baseline: Normal | 6
  Baseline: Abnormal NCS | 2
  Baseline: Abnormal CS | 0
  Week 26: number analyzed (Participants) | 9
  Week 26: Normal | 6
  Week 26: Abnormal NCS | 3
  Week 26: Abnormal CS | 0
  Week 52: number analyzed (Participants) | 7
  Week 52: Normal | 5
  Week 52: Abnormal NCS | 2
  Week 52: Abnormal CS | 0
  Week 104: number analyzed (Participants) | 7
  Week 104: Normal | 4
  Week 104: Abnormal NCS | 3
  Week 104: Abnormal CS | 0
  Week 156: number analyzed (Participants) | 7
  Week 156: Normal | 5
  Week 156: Abnormal NCS | 2
  Week 156: Abnormal CS | 0

36. Secondary Outcome: Number of Participants in Categories of Brain Magnetic Resonance Imaging (MRI) Results at Baseline and Weeks 26, and 156
Description: All continuous MRI variables were summarized using descriptive statistics for each visit. The overall interpretation of the readings were summarized in 2 categories as: normal, and abnormal. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants
  Baseline: number analyzed (Participants) | 10
  Baseline: Normal | 6
  Baseline: Abnormal | 4
  Week 26: number analyzed (Participants) | 9
  Week 26: Normal | 7
  Week 26: Abnormal | 2
  Week 156: number analyzed (Participants) | 7
  Week 156: Normal | 4
  Week 156: Abnormal | 3

37. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Weeks 26, 52, 104, and 156
Description: Estimated glomerular filtration rate was used to measure level of kidney function and determine the stage of kidney disease. Change from baseline in eGFR was obtained by subtracting baseline value from post-baseline value at Weeks 26, 52, 104 and 156. For this analysis, baseline was defined as initial ACT13739 study baseline.
Time Frame: Baseline of ACT13739 study and Weeks 26, 52, 104, and 156 post-ACT13739 baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
mL/min/1.73m^2
  Week 26: number analyzed (Participants) | 7
  Week 26 | -3.43 (8.64)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -5.57 (11.07)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -5.71 (10.23)
  Week 156: number analyzed (Participants) | 6
  Week 156 | -4.83 (17.54)

38. Secondary Outcome: Chitotriosidase (Chit1) Plasma Concentration Levels at Weeks 52, 104,156 and 160 (End of Treatment Follow-up)
Description: Plasma concentrations of Chit1 over time were determined using mass spectrometry (MS)-based assay. For the analysis, 52 ng/mL was considered as the lower limit of quantification. Although identified in protocol as a secondary endpoint, plasma Chit1 is also an exploratory measure. Only LTS14116 timepoints were analyzed and are presented. Data summarized are the measured values at each time point (not change from baseline). Here, measured value '0.000' denotes no chitotriosidase detected in plasma for the 5 participants at Week 156 reported by laboratory for all evaluable participants.
Time Frame: Weeks 52, 104, 156 and 160 (End of Treatment Follow-up) post-ACT13739 baseline
Population: Analysis population included participants in LTS14116 study with evaluable plasma Chit1 data. Only data collected during LTS14116 study were included in analysis. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 7
ng/mL
  Week 52 | 35.965 (46.520)
  Week 104 | 12.785 (20.993)
  Week 156: number analyzed (Participants) | 5
  Week 156 | 0.000 (0.000)
  Week 160 (End of Treatment Follow-up): number analyzed (Participants) | 4
  Week 160 (End of Treatment Follow-up) | 6.483 (6.309)

ADVERSE EVENTS:
Time Frame: From baseline of ACT13739 study up to 37 months post-ACT13739 baseline.
Description: Reported AEs were TEAEs, defined as AEs that developed/worsened during TEAE period (period from the first administration of study drug in ACT13739 through the last administration of the study drug in the combined ACT13739/LTS14116 treatment period plus 1 month or end of study participation for participant, whichever occurs first). Analysis was performed on safety population.
Arm/Group | GZ/SAR402671
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GZ/SAR402671 (N=11)
Haemolysis (Blood and lymphatic system disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Floppy infant (Musculoskeletal and connective tissue disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GZ/SAR402671 (N=11)
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Vertigo (Ear and labyrinth disorders) | 1
Blepharitis (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Lenticular opacities (Eye disorders) | 1
Retinal vascular disorder (Eye disorders) | 2
Vision blurred (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Oesophageal discomfort (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Feeling hot (General disorders) | 2
Influenza like illness (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Temperature intolerance (General disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 2
Tooth fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 1
Vibration test abnormal (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Amnesia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Hemiparesis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
White matter lesion (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Micturition frequency decreased (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Angiokeratoma (Skin and subcutaneous tissue disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT02489344/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02489344/SAP_001.pdf